CLINICAL TRIAL: NCT02311699
Title: Using Cultural Ceremonies to Reduce Intimate Partner Violence and HIV Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Ethiopian Public Health Association (Unknown); Addis Ababa University (Other); EngenderHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALJameelPAL
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: HIV
Keywords: Gender; Physical Violence; Sexual Violence; HIV; AIDS; Prevention; Community Intervention; Ethiopia; Intimate Partner Violence
MeSH Terms: conditions — Coitus; Acquired Immunodeficiency Syndrome | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Women Only (Experimental): Groups of women will receive the behavioral intervention to reduce IPV and HIV. Sessions will be led by female facilitators.
  Interventions: Behavioral: Intervention to reduce IPV and HIV
- Men Only (Experimental): Groups of men will receive the behavioral intervention to reduce IPV and HIV. Sessions will be led by male facilitators.
  Interventions: Behavioral: Intervention to reduce IPV and HIV
- Couples (Experimental): Couples will receive the behavioural intervention to reduce IPV and HIV. Sessions will be led by a male and a female facilitator.
  Interventions: Behavioral: Intervention to reduce IPV and HIV
- Control Group (No Intervention): Community members in the control villages will receive a short informational session on violence reduction.

INTERVENTIONS:
Behavioral: Intervention to reduce IPV and HIV — The Ethiopian traditional coffee ceremony will be used as an entry point for a community based intervention to provide information, change behaviour around IPV and improve gender equity and intra-couple relations. The coffee ceremony is a culturally established forum for community discussion and conflict resolution and an integral part of Ethiopian life. The intervention will involve regular coffee ceremonies, during which approximately 20 members of the community will participate in education and discussions centred on gender issues, sexuality, communication and conflict resolution, HIV/AIDS and its link with violence, as well as HIV/AIDS prevention. Each coffee ceremony will be moderated by a female or male facilitator trained in participatory learning, moderation, HIV/AIDS prevention, counselling, and gender issues. The intervention will involve 14 two-hour session per group of participants.
  Arms: Couples; Men Only; Women Only

SUMMARY:
Violence against women (VAW), the most extreme manifestation of the unequal power balance between women and men, is a major global public health concern. One of the most common forms of VAW is that perpetrated by a husband or other intimate partner. In Ethiopia, 70.9% of women reported having experienced physical and/or sexual intimate partner violence (IPV) in their lifetime, demonstrating the pervasiveness of the problem. A growing body of evidence has also linked IPV and HIV risk.

This study is a cluster randomized controlled trial assessing the impact of a community-based intervention focused on Intimate Partner Violence and HIV delivered in the context of the Ethiopian coffee ceremony, a culturally established forum for community discussion and conflict resolution. Villages will be randomly assigned to one of 4 study arms (3 intervention and one control arm): 1) Women only participate in the intervention, 2) Men only participate, 3) Both men and women (couples) participate, 4) Women and men receive the control intervention comprising a short informational session on violence reduction.

ELIGIBILITY:
Inclusion Criteria:

* currently married or cohabitating with partner
* residing in selected village for at least 6 months

Exclusion Criteria:

* eligible women who do not consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6800 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Experience of physical violence by an intimate partner in the previous 12 months (among married or co-habitating women) | 12 months
Experience of sexual violence by an intimate partner in the previous 12 months (among married or co-habitating women) | 12 months

SECONDARY OUTCOMES:
Perpetration of physical violence towards an intimate partner in previous 12 months (among married or co-habitating men) | 12 months
Perpetration of sexual violence towards an intimate partner in previous 12 months (among married or co-habitating men) | 12 months
Proportion with comprehensive HIV/AIDS knowledge (among married or co-habitating men or women) | 18 months
Proportion using a condom at last high risk sexual intercourse (among married or co-habitating men or women) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Sharma, MD, MPH, Principal Investigator — Massachusetts Institute of Technology; Jessica Leight, PhD, Principal Investigator — Williams College; Negussie Deyessa, PhD, Principal Investigator — Addis Ababa University
Locations (1):
- Ethiopian Public Health Association, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Leight J, Deyessa N, Sharma V. Cost-effectiveness analysis of an intimate partner violence prevention intervention targeting men, women and couples in rural Ethiopia: evidence from the Unite for a Better Life randomised controlled trial. BMJ Open. 2021 Mar 29;11(3):e042365. doi: 10.1136/bmjopen-2020-042365. PMID 33782020
- [Derived] Leight J, Deyessa N, Verani F, Tewolde S, Sharma V. Community-level spillover effects of an intervention to prevent intimate partner violence and HIV transmission in rural Ethiopia. BMJ Glob Health. 2021 Jan;6(1):e004075. doi: 10.1136/bmjgh-2020-004075. PMID 33509840
- [Derived] Leight J, Deyessa N, Verani F, Tewolde S, Sharma V. An intimate partner violence prevention intervention for men, women, and couples in Ethiopia: Additional findings on substance use and depressive symptoms from a cluster-randomized controlled trial. PLoS Med. 2020 Aug 18;17(8):e1003131. doi: 10.1371/journal.pmed.1003131. eCollection 2020 Aug. PMID 32810147
- [Derived] Sharma V, Leight J, Verani F, Tewolde S, Deyessa N. Effectiveness of a culturally appropriate intervention to prevent intimate partner violence and HIV transmission among men, women, and couples in rural Ethiopia: Findings from a cluster-randomized controlled trial. PLoS Med. 2020 Aug 18;17(8):e1003274. doi: 10.1371/journal.pmed.1003274. eCollection 2020 Aug. PMID 32810146